CLINICAL TRIAL: NCT05631405
Title: Efficacy of Dengue Infection With Warning Signs Treated With Dexamethasone
Brief Title: Efficacy of Dengue Infection With Warning Signs Treated With Dexamethasone (DengDex Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Principal investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB.436/65
Record Dates: First submitted 2022-11-09; First posted 2022-11-30 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Severe Dengue
Keywords: Severe Dengue; Dexamethasone; Steroid
MeSH Terms: conditions — Severe Dengue | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Intervention (Experimental)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Patients treated with dexamethasone
  Arms: Intervention
Drug: Placebo — Patients treated with placebo
  Arms: Placebo

SUMMARY:
The goal of this randomized double-blinded placebo-controlled trial is to learn about dexamethasone and the treatment of severe dengue population. The main question it aims to answer are steroid therapy may be effective in dengue.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed Dengue infected patients (Positive NS1 Ag or anti-DENV IgM by Dengue Duo test)
* And still in febrile phase (Body temp>37.5 C)
* Shock : Sys<90mmHg or Narrow PP (<20mmHg) orTachycardia (pulse>100/min) with Hematocrit decreased ≥20 %
* Fluid accumulation and respiratory distress
* Severe bleeding
* Severe organ involvement

Exclusion Criteria:

* Severe dengue> 24 hrs
* Dengue without warning signs
* Pregnancy
* Patient who receieved any steroid within 1 week

Ages: 7 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days
  The use of steroids in dengue will reduce mortality in rate

SECONDARY OUTCOMES:
Length of hospital stay | 28 days
  The use of steroids in dengue will reduce Length of hospital stay in day

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Chulalongkorn University, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No